CLINICAL TRIAL: NCT05017012
Title: A Phase 1 Clinical Study to Evaluate the Bioavailability of Pembrolizumab Via Subcutaneous Injection of MK-3475A, a Formulation of Pembrolizumab With MK-5180, in Participants With Advanced Solid Tumors
Brief Title: A Study to Evaluate the Bioavailability of Pembrolizumab (MK-3475) Via Subcutaneous (SC) Injection of Pembrolizumab Formulated With Berahyaluronidase Alfa (MK-5180) [MK-3475A] In Advanced Solid Tumors (MK-3475A-C18)
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 3475A-C18; MK-3475A-C18 (Other: MSD); jRCT2031220507 (Registry Identifier: Japan Registry of Clinical Trials (jRCT)); 2023-505340-19-00 (Registry Identifier: EU CT); U1111-1291-5232 (Registry Identifier: UTN); 2021-001569-18 (EudraCT Number)
Record Dates: First submitted 2021-08-18; First posted 2021-08-23 (Actual); Last update posted 2026-01-08 (Actual); Status verified 2025-12

CONDITIONS: Advanced or Metastatic Solid Tumors
Keywords: Programmed Cell Death-1 (PD1, PD-1); Programmed Death-Ligand 1 (PDL1, PD-L1)
MeSH Terms: conditions — Parkinson Disease 4, Autosomal Dominant Lewy Body | interventions — pembrolizumab; Pemetrexed; Carboplatin; Paclitaxel; 130-nm albumin-bound paclitaxel; Albumin-Bound Paclitaxel; Axitinib; Cisplatin

STUDY DESIGN:
Masking Description: None (Open-label)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Pembrolizumab Conc1 [dose 1]/Berahyaluronidase alfa (Experimental): Participants receive pembrolizumab (+) berahyaluronidase alfa (pembrolizumab Conc1 [dose 1] + berahyaluronidase alfa) SC on Day 1 of Cycles 1 and 3 plus 400 mg pembrolizumab intravenously (IV) on Day 1 of Cycles 2 and 4 to 18, with or without background standard of care (SOC) chemotherapy as appropriate for the indication. A cycle is 42 days.
  Interventions: Biological: Pembrolizumab (+) Berahyaluronidase alfa; Biological: Pembrolizumab; Drug: Pemetrexed; Drug: Carboplatin; Drug: Paclitaxel; Drug: Nab-paclitaxel; Drug: Axitinib; Drug: Cisplatin
- Pembrolizumab Conc2 [dose 1]/Berahyaluronidase alfa (Experimental): Participants receive pembrolizumab (+) berahyaluronidase alfa (pembrolizumab Conc2 [dose 1] + Berahyaluronidase alfa) SC on Day 1 of Cycles 1 and 3 plus 400 mg pembrolizumab IV on Day 1 of Cycles 2 and 4 to 18, with or without background SOC chemotherapy as appropriate for the indication. A cycle is 42 days.
  Interventions: Biological: Pembrolizumab (+) Berahyaluronidase alfa; Biological: Pembrolizumab; Drug: Pemetrexed; Drug: Carboplatin; Drug: Paclitaxel; Drug: Nab-paclitaxel; Drug: Axitinib; Drug: Cisplatin
- Pembrolizumab Conc1 [dose 1]/Berahyaluronidase alfa + SOC Chemotherapy (Experimental): Participants in Japan receive pembrolizumab (+) berahyaluronidase alfa (pembrolizumab Conc1 [dose 1] + berahyaluronidase alfa) SC on Day 1 of Cycle 1, with background SOC chemotherapy, and then receive 400 mg pembrolizumab IV on Day 1 of Cycles 2 to 18, with background SOC chemotherapy. A cycle is 42 days.
  Interventions: Biological: Pembrolizumab (+) Berahyaluronidase alfa; Biological: Pembrolizumab; Drug: Pemetrexed; Drug: Carboplatin; Drug: Paclitaxel; Drug: Nab-paclitaxel; Drug: Cisplatin
- Pembrolizumab Conc1 [dose 2]/Berahyaluronidase alfa (Experimental): Participants receive pembrolizumab (+) berahyaluronidase alfa (pembrolizumab Conc1 [dose 2] + berahyaluronidase alfa) SC on Day 1 of Cycles 1 to 35 without background standard of care (SOC) chemotherapy. A cycle is 21 days.
  Interventions: Biological: Pembrolizumab (+) Berahyaluronidase alfa

INTERVENTIONS:
Biological: Pembrolizumab (+) Berahyaluronidase alfa — Pembrolizumab (+) Berahyaluronidase alfa is a fixed-dose formulation of pembrolizumab (either Conc1 or Conc2) and berahyaluronidase alfa for SC administration.
  Other Names: MK-3475A
Biological: Pembrolizumab — Participants will receive pembrolizumab 400 mg IV.
  Other Names: Keytruda; MK-3475
  Arms: Pembrolizumab Conc1 [dose 1]/Berahyaluronidase alfa; Pembrolizumab Conc1 [dose 1]/Berahyaluronidase alfa + SOC Chemotherapy; Pembrolizumab Conc2 [dose 1]/Berahyaluronidase alfa
Drug: Pemetrexed — Participants may receive 500 mg/m^2 IV every 3 weeks (Q3W) Day 1 and Day 22 of Cycles 1 to 18 as background SOC treatment during the study, as applicable to their diagnosis.
  Other Names: Alimta
  Arms: Pembrolizumab Conc1 [dose 1]/Berahyaluronidase alfa; Pembrolizumab Conc1 [dose 1]/Berahyaluronidase alfa + SOC Chemotherapy; Pembrolizumab Conc2 [dose 1]/Berahyaluronidase alfa
Drug: Carboplatin — Participants may receive 5 mg/mL/min IV (nonsquamous) or 6 mg/mL/min IV (squamous) on Day 1 of each 21-day cycle for 4 cycles as background SOC treatment during the study, as applicable to their diagnosis.
  Arms: Pembrolizumab Conc1 [dose 1]/Berahyaluronidase alfa; Pembrolizumab Conc1 [dose 1]/Berahyaluronidase alfa + SOC Chemotherapy; Pembrolizumab Conc2 [dose 1]/Berahyaluronidase alfa
Drug: Paclitaxel — Participants may receive 200 mg/m^2 IV on Day 1 of each 21-day cycle for 4 cycles as background SOC treatment during the study, as applicable to their diagnosis.
  Other Names: Taxol
  Arms: Pembrolizumab Conc1 [dose 1]/Berahyaluronidase alfa; Pembrolizumab Conc1 [dose 1]/Berahyaluronidase alfa + SOC Chemotherapy; Pembrolizumab Conc2 [dose 1]/Berahyaluronidase alfa
Drug: Nab-paclitaxel — Participants may receive 100 mg/m2 IV on Day 1, 8, and 15 of each 21-day cycle for 4 cycles as background SOC treatment during the study, as applicable to their diagnosis.
  Other Names: Albumin-bound paclitaxel
  Arms: Pembrolizumab Conc1 [dose 1]/Berahyaluronidase alfa; Pembrolizumab Conc1 [dose 1]/Berahyaluronidase alfa + SOC Chemotherapy; Pembrolizumab Conc2 [dose 1]/Berahyaluronidase alfa
Drug: Axitinib — Participants may receive 5 mg orally twice daily continuously as background SOC treatment during the study, as applicable to their diagnosis.
  Arms: Pembrolizumab Conc1 [dose 1]/Berahyaluronidase alfa; Pembrolizumab Conc2 [dose 1]/Berahyaluronidase alfa
Drug: Cisplatin — Participants may receive 75 mg/m^2 IV on Day 1 of each 21-day cycle for 4 cycles as background SOC treatment during the study, as applicable to their diagnosis.
  Other Names: Platinol-AQ
  Arms: Pembrolizumab Conc1 [dose 1]/Berahyaluronidase alfa; Pembrolizumab Conc1 [dose 1]/Berahyaluronidase alfa + SOC Chemotherapy; Pembrolizumab Conc2 [dose 1]/Berahyaluronidase alfa

SUMMARY:
This is a study to assess the pharmacokinetics, safety, and tolerability of pembrolizumab formulated with berahyaluronidase when administered as a SC injection to participants with advanced solid tumors. Participants will receive SC injections of pembrolizumab (+) berahyaluronidase alfa containing one of 2 different concentrations (Conc) of pembrolizumab, Conc1 and Conc2, corresponding to a pembrolizumab dose level of dose 1 for Arms 1, 2, and 3 and dose 2 for Arm 4.

ELIGIBILITY:
Inclusion Criteria:

* Has a histologically- or cytologically-confirmed advanced/metastatic solid tumor.
* Can provide archival tumor tissue sample or newly obtained core or excisional biopsy of a tumor lesion not previously irradiated.
* Has a measurable disease per Response Evaluation Criteria in Solid Tumors (RECIST) 1.1.
* Has a performance status of 0 or 1 on the Eastern Cooperative Oncology Group Performance Scale.
* Demonstrates adequate organ function.

Exclusion Criteria:

* Has a diagnosis of immunodeficiency or is receiving chronic systemic steroid therapy (in dosing exceeding 10 mg daily of prednisone equivalent) or any other form of immunosuppressive therapy within 7 days prior to the first dose of study medication.
* Has had chemotherapy, definitive radiation, or biological cancer therapy within 4 weeks (2 weeks for palliative radiation) before the first dose of study intervention, or has not recovered to National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) Grade 1 or better from any adverse events (AEs) that were due to cancer therapeutics administered more than 4 weeks earlier (this includes participants with previous immunomodulatory therapy with residual immune-related AEs).
* Has a history of a second malignancy, unless potentially curative treatment has been completed with no evidence of malignancy for 2 years
* Has clinically active central nervous system (CNS) metastases and/or carcinomatous meningitis.
* Has severe hypersensitivity (≥Grade 3) to pembrolizumab and/or any of its excipients.
* Has an active infection requiring therapy.
* Has a history of (noninfectious) pneumonitis/interstitial lung disease that required steroids or current pneumonitis/interstitial lung disease.
* Has an active autoimmune disease that has required systemic treatment in the past 2 years.
* Has known hepatitis B or C infections or known to be positive for hepatitis B surface antigen (HBsAg)/hepatitis B virus deoxyribonucleic acid (DNA) or hepatitis C antibody and ribonucleic acid (RNA)
* Human immunodeficiency virus (HIV)-infected participants with a history of Kaposi's sarcoma and/or Multicentric Castleman's Disease.
* Has a history or current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the study, interfere with the participant's participation for the full duration of the study, or is not in the best interest of the participant to participate, in the opinion of the treating investigator.
* Is pregnant, breastfeeding, or expecting to conceive or father children within the projected duration of the study.
* Has not fully recovered from any effects of major surgery without significant detectable infection.
* Has symptomatic ascites or pleural effusion.
* Has preexisting peripheral neuropathy that is >Grade 2 by latest NCI CTCAE version 5.
* Has a known sensitivity to recombinant hyaluronidase or other form of hyaluronidase.
* Has a history of severe hypersensitivity reaction (eg, generalized rash/erythema, hypotension, bronchospasm, angioedema, or anaphylaxis) to pemetrexed, cisplatin, axitinib, carboplatin, paclitaxel, or nab-paclitaxel.
* Has received a live or live-attenuated vaccine within 30 days before the first dose of study intervention.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Estimated)
Dates: Start 2021-09-21 (Actual); Primary Completion 2026-05-11 (Estimated); Study Completion 2026-05-11 (Estimated)

PRIMARY OUTCOMES:
Arms 1, 2, and 3: Pembrolizumab Trough Concentration (Ctrough) After pembrolizumab (+) berahyaluronidase alfa Treatment | Predose (0-3 hours) and postdose (0-10 minutes) on Cycle 1 Day 1; any time on Cycle 1 Days 2, 3, 4, 5, 6, 8, 10, 15, 22, 29, and 36. Cycle = 42 days
  Ctrough is defined as the observed trough concentration measured during the absorption phase, prior to SC injection of pembrolizumab (+) berahyaluronidase alfa. Ctrough will be reported for Arms 1, 2, and 3.
Arms 1, 2, and 3: Pembrolizumab Maximum Plasma Concentration (Cmax) After pembrolizumab (+) berahyaluronidase alfa Treatment | Predose (0-3 hours) and postdose (0-10 minutes) on Cycle 1 Day 1; any time on Cycle 1 Days 2, 3, 4, 5, 6, 8, 10, 15, 22, 29, and 36. Cycle = 42 days
  Cmax is defined as the maximum plasma concentration measured during the absorption phase, following SC injection of pembrolizumab (+) berahyaluronidase alfa. Cmax will be reported for Arms 1, 2, and 3.
Arms 1, 2, and 3: Pembrolizumab Time of Maximum Plasma Concentration (Tmax) After pembrolizumab (+) berahyaluronidase alfa Treatment | Predose (0-3 hours) and postdose (0-10 minutes) on Cycle 1 Day 1; any time on Cycle 1 Days 2, 3, 4, 5, 6, 8, 10, 15, 22, 29, and 36. Cycle = 42 days
  Tmax is defined as the time to maximum plasma concentration measured during the absorption phase, following SC injection of pembrolizumab (+) berahyaluronidase alfa. Tmax will be reported for Arms 1, 2, and 3.
Arms 1, 2, and 3: Pembrolizumab Area under the Curve (AUC) After pembrolizumab (+) berahyaluronidase alfa Treatment | Predose (0-3 hours) and postdose (0-10 minutes) on Cycle 1 Day 1; any time on Cycle 1 Days 2, 3, 4, 5, 6, 8, 10, 15, 22, 29, and 36. Cycle = 42 days
  AUC is defined as the area under the curve measured during the absorption phase, following SC injection of pembrolizumab (+) berahyaluronidase alfa. AUC will be reported for Arms 1, 2, and 3.
Arms 1 and 2: Pembrolizumab Bioavailability (F) After pembrolizumab (+) berahyaluronidase alfa Treatment | At designated timepoints in Cycles 1 to 4 (up to 127 days). Cycle = 42 days
  Bioavailability (F) is defined as the percentage (or the fraction F) of an administered SC dose that reaches the systemic circulation unaltered during the absorption phase, following SC injection of pembrolizumab (+) berahyaluronidase alfa. F will be reported for Arms 1 and 2.
Arm 3 (Japan): Number of Participants Who Experience a Dose-Limiting Toxicity (DLT) | Up to 21 days of Cycle 1 (each cycle is 42 days)
  DLT is defined as any of the following toxicities, if assessed by the investigator to be related to study treatment: Grade (Gr) 4 nonhematologic toxicity (not laboratory); Gr 4 hematologic toxicity lasting ≥7 days, except thrombocytopenia: Gr 4 thrombocytopenia of any duration; Gr 3 thrombocytopenia associated with clinically significant bleeding; thrombocytopenia requiring platelet transfusion; anemia requiring red blood cell transfusion; Nonhematologic AE Gr ≥3 in severity, with exceptions; Any Gr 3 or 4 nonhematologic laboratory abnormality if: clinically significant medical intervention is required, or if abnormality leads to hospitalization, persists for >1 week or results in drug-induced liver injury with exceptions; Gr 3 or Gr 4 febrile neutropenia; Prolonged delay (>2 weeks) during Cycle 1 Days 1 to 21 due to treatment-related toxicity; Treatment-related toxicity resulting in participant study treatment discontinuation during Cycle 1 Days 1 to 21; Gr 5 toxicity.
Arm 3 (Japan): Number of Participants with Adverse Events (AEs) | Up to approximately 120 weeks
  An AE is any untoward medical occurrence in a clinical study participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention. The number of participants with an AE will be reported for Arm 3.
Arm 3 (Japan): Number of Participants who Discontinue Study Treatment Due to an AE | Up to approximately 108 weeks
  An AE is any untoward medical occurrence in a clinical study participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention. The number of participants who discontinue study treatment due to an AE will be reported for Arm 3.
Arm 3 (Japan): Number of Participants with Injection Site Signs and Symptoms as Assessed by the Subcutaneous Injection Site Signs and Symptoms Questionnaire | Day 1 of Cycle 1: Up to 60 minutes postdose. Cycle = 42 days
  Approximately 60 minutes post injection of pembrolizumab (+) berahyaluronidase alfa on Day 1 of Cycles 1 and 3, participants are to complete the Subcutaneous Injection Site Signs and Symptoms Questionnaire. Participants are asked to rate any pain, itching, swelling and redness they experience at the pembrolizumab SC injection site from "None" to "Severe". The number of participants who experience an injection site sign or symptom will be reported for Arm 3.
Arm 4: Pembrolizumab Trough Concentration (Ctrough) After pembrolizumab (+) berahyaluronidase alfa Treatment | Predose (0-3 hours) on Day 1 of Cycles 1 and 6; any time on Days 2, 4, 6, 10, and 15 of Cycles 1 and 6. Cycle = 21 days
  Ctrough is defined as the observed trough concentration measured during the absorption phase, prior to SC injection of pembrolizumab (+) berahyaluronidase alfa. Ctrough will be reported for Arm 4.
Arm 4: Pembrolizumab Maximum Plasma Concentration (Cmax) After pembrolizumab (+) berahyaluronidase alfa Treatment | Predose (0-3 hours) on Day 1 of Cycles 1 and 6; any time on Days 2, 4, 6, 10, and 15 of Cycles 1 and 6. Cycle = 21 days
  Cmax is defined as the maximum plasma concentration measured during the absorption phase, following SC injection of pembrolizumab (+) berahyaluronidase alfa. Cmax will be reported for Arm 4.
Arm 4: Pembrolizumab Area under the Curve (AUC) After pembrolizumab (+) berahyaluronidase alfa Treatment | Predose (0-3 hours) on Day 1 of Cycles 1 and 6; any time on Days 2, 4, 6, 10, and 15 of Cycles 1 and 6. Cycle = 21 days
  AUC is defined as the area under the curve measured during the absorption phase, following SC injection of pembrolizumab (+) berahyaluronidase alfa. AUC will be reported for Arm 4.

SECONDARY OUTCOMES:
Number of Participants Positive for Anti-Pembrolizumab Antibodies After pembrolizumab (+) berahyaluronidase alfa Treatment | Predose (0-3 hours) on Day 1 of Cycles 1 and 3. Cycle = 42 days.
  Blood samples are to be collected at designated time points for the determination of the presence or absence of anti-pembrolizumab antibodies. The percentage of participants who develop anti-pembrolizumab antibodies will be reported.
Arms 1, 2, and 4: Number of Participants with Adverse Events (AEs) | Up to approximately 120 weeks
  An AE is any untoward medical occurrence in a clinical study participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention. The number of participants with an AE will be reported for Arms 1, 2, and 4.
Arms 1, 2, and 4: Number of Participants who Discontinue Study Treatment Due to an AE | Up to approximately 108 weeks
  An AE is any untoward medical occurrence in a clinical study participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention. The number of participants who discontinue study treatment due to an AE will be reported for Arms 1, 2, and 4.
Arms 1 and 2: Number of Participants with Injection Site Signs and Symptoms as Assessed by the Subcutaneous Injection Site Signs and Symptoms Questionnaire | Day 1 of Cycles 1 and 3: Up to 60 minutes postdose. Cycle = 42 days.
  Approximately 60 minutes post injection of pembrolizumab (+) berahyaluronidase alfa on Day 1 of Cycles 1 and 3, participants are to complete the Subcutaneous Injection Site Signs and Symptoms Questionnaire. Participants are asked to rate any pain, itching, swelling and redness they experience at the pembrolizumab SC injection site from "None" to "Severe". The number of participants who experience an injection site sign or symptom will be reported for Arms 1 and 2.
Arm 4: Number of Participants with Injection Site Signs and Symptoms as Assessed by the Subcutaneous Injection Site Signs and Symptoms Questionnaire | Cycle 1 Day 1: Up to 60 minutes postdose. Cycle = 21 days
  Approximately 60 minutes post injection of pembrolizumab (+) berahyaluronidase alfa on Day 1 of Cycle 1, participants are to complete the Subcutaneous Injection Site Signs and Symptoms Questionnaire. Participants are asked to rate any pain, itching, swelling and redness they experience at the pembrolizumab SC injection site from "None" to "Severe". The number of participants who experience an injection site sign or symptom will be reported for Arm 4.
Arm 3 (Japan): Pembrolizumab Bioavailability (F) After pembrolizumab (+) berahyaluronidase alfa Treatment | At designated timepoints in Cycles 1-2 (up to 84 days). Cycle = 42 days
  Bioavailability (F) is defined as the percentage (or the fraction F) of an administered SC dose that reaches the systemic circulation unaltered during the absorption phase, following SC injection of pembrolizumab (+) berahyaluronidase alfa. F will be reported for Arm 3.

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC
Locations (22):
- Chile (3):
  - FALP-UIDO ( Site 0101), Santiago, Region M. de Santiago
  - Bradfordhill ( Site 0100), Santiago, Region M. de Santiago
  - James Lind Centro de Investigación del Cáncer ( Site 0102), Temuco, Región de la Araucanía
- Hungary (2):
  - Országos Onkológiai Intézet-Urogenital Tumors Department and Clinical Pharmacology ( Site 0021), Budapest, Pest County
  - Magyar Honvedseg Egeszsegugyi Kozpont-Onkologiai Osztaly ( Site 0020), Budapest
- Japan (5):
  - Kansai Medical University Hospital ( Site 0112), Hirakata, Osaka
  - Saitama Prefectural Cancer Center ( Site 0110), Ina-machi, Saitama
  - Shizuoka Cancer Center ( Site 0111), Nagaizumi-cho,Sunto-gun, Shizuoka
  - National Hospital Organization Kyushu Cancer Center ( Site 0114), Fukuoka
  - Osaka International Cancer Institute ( Site 0113), Osaka
- South Africa (7):
  - CANCERCARE LANGENHOVEN DRIVE ONCOLOGY CENTRE ( Site 0051), Port Elizabeth, Eastern Cape
  - Medical Oncology Centre of Rosebank ( Site 0058), Johannesburg, Gauteng
  - Steve Biko Academic Hospital-Medical Oncology ( Site 0057), Pretoria, Gauteng
  - LIFE GROENKLOOF-Mary Potter Cancer Centre ( Site 0052), Pretoria, Gauteng
  - Sandton Oncology Medical Group (Pty) Ltd-Research ( Site 0053), Sandton, Gauteng
  - Cape Town Oncology Trials ( Site 0050), Cape Town, Western Cape
  - Cancercare Rondebosch Oncology-Clinical trials ( Site 0055), Rondebosch, Western Cape
- South Korea (2):
  - Severance Hospital, Yonsei University Health System ( Site 0062), Seoul
  - Samsung Medical Center ( Site 0063), Seoul
- Spain (3):
  - Hospital Universitario Virgen de la Victoria-Phase I Trials Unit ( Site 0042), Málaga, Andalusia
  - HOSPITAL CLÍNIC DE BARCELONA-Department of Medical Oncology ( Site 0043), Barcelona, Catalonia
  - HOSPITAL GENERAL UNIVERSITARIO GREGORIO MARAÑON-ONCOLOGY ( Site 0040), Madrid, Madrid, Comunidad de

IPD SHARING:
Plan to Share IPD: Yes
https://trialstransparency.msdclinicaltrials.com/pdf/ProcedureAccessClinicalTrialData.pdf
URL: https://externaldatasharing-msd.com/

REFERENCES:
- [Derived] Cohen GL, Coetzee C, Walton CA, Reig Torras O, Chul Cho B, McAdam G, Rojas CI, Medina Rodriguez L, Papai Z, Chan SW, Rapoport BL, Caglevic C, Yanez Weber P, Takahashi T, Kurata T, Song G, Cohen JW, Akala OO, Khanyile R. Pharmacokinetics and bioavailability of pembrolizumab with berahyaluronidase alfa for subcutaneous administration in participants with advanced or metastatic solid tumors: The phase 1 study 3475A-C18. Eur J Cancer. 2025 Nov 17;230:115709. doi: 10.1016/j.ejca.2025.115709. Epub 2025 Aug 9. PMID 40957773
- See also: Merck Clinical Trials Information — http://merckclinicaltrials.com
- See also: Plain Language Summary — https://msd.trialsummaries.com/Study/StudyDetails?id=26240&tenant=MT_MSD_9011